CLINICAL TRIAL: NCT03696745
Title: The Treatment of Premature Infants With Brain Injury by Autologous Umbilical Cord Blood Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yangjie, Professor, Guangdong Women and Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangdongW C H
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Safety Issues; Effect of Drugs
Keywords: Autologous Umbilical Cord Blood Stem Cells; Safety; Effect; brain injury
MeSH Terms: conditions — Brain Injuries | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): preterm infants with severe hypoxic ischemic encephalopathy receive only 0.9% Sodium-chloride
  Interventions: Drug: 0.9% Sodium-chloride
- infusion (Experimental): preterm infants with severe hypoxic ischemic encephalopathy will receive up to 4 infusions of their own volume reduced cord blood stem cells. The number of doses will be determined by the amount of available cord blood stem cells. The dose for each infusion is 5x107 cells/kg
  Interventions: Other: autologous umbilical cord blood stem cells

INTERVENTIONS:
Other: autologous umbilical cord blood stem cells — autologous umbilical cord blood stem cells treatment for brain injury for safety and effect evaluation
  Arms: infusion
Drug: 0.9% Sodium-chloride — 0.9% Sodium-chloride in control group
  Arms: Placebo

SUMMARY:
To study the safety and effect of autologous umbilical cord blood stem cells for treatment brain injury

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effect of infusions of autologous (the patient's own)umbilical cord blood stem cells in newborn infants with hypoxic-ischemic encephalopathy. For this study, infants who have signs of moderate to severe encephalopathy at birth whose mothers have previously consented to providing cord blood stem cells for the Gunagdong Cord Blood Bank,or provided verbal consent for cord blood collection for the possibility of their baby's participation in this trial, can receive their own cord blood stem cells if an adequate number of cells that meet Guangdong Cord Blood Bank Quality standards are available in the first 14 postnatal days. Study activities also include serial blood draws concurrent with clinically indicated blood draws with a total volume of no more than 5 milliliters (1 teaspoon) from all study related tests. Babies will be followed for neurodevelopmental outcome at 4 - 6 and 9 - 12 months. MRI's will be obtained per clinical routine and results will be analyzed and described in study reports.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must have consented for cord blood collection at delivery
* cord blood must be available for extraction of stem cells.

  ->28 weeks gestation,<37weeks gestation
* cord or neonatal pH<7.0 or base deficit>16 milliequivalents per liter (mEq/L) or history of acute perinatal event
* either a 10 minute Apgar < 5 or continued need for ventilation.
* All infants must have signs of encephalopathy within 6 hours of age.

Exclusion Criteria:

* Presence of known chromosomal anomaly.
* Presence of major congenital anomalies.
* Severe intrauterine growth restriction (weight <1800g)
* Infants in extremis for whom no additional intensive therapy will be offered by attending neonatologist.
* Parents refuse consent.
* Attending neonatologist refuses consent.
* Failure to collect the infant's cord blood and/or laboratory unable to process cord blood.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
safety of autologous umbilical cord blood stem cells infusion in enrolled preterm infants | during infusion 24 hours after infusion
  Adverse event rates occurring will be compared between the autologous umbilical cord blood stem cells recipients and control group

SECONDARY OUTCOMES:
effect of autologous umbilical cord blood stem cells infusion in enrolled preterm infants | 1 year
  the effect of autologous umbilical cord blood stem cells infusion will be measured by neurodevelopmental function at 4 - 6 months and 9 - 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PHD, Principal Investigator — Gunagzhou,Guangdong,China,511442

IPD SHARING:
Plan to Share IPD: Undecided